CLINICAL TRIAL: NCT02344355
Title: Pharmacological Ascorbate Combined With Radiation and Temozolomide in Glioblastoma Multiforme: A Phase 2 Trial
Brief Title: A Phase 2 Trial of High-Dose Ascorbate in Glioblastoma Multiforme
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bryan Allen (Other)
Collaborators: Holden Comprehensive Cancer Center (Other); National Cancer Institute (NCI) (NIH); Gateway for Cancer Research (Other)
Responsible Party: Sponsor-Investigator, Bryan Allen, Assistant Professor, Radiation Oncology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201504786
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma Multiforme
Keywords: Ascorbic Acid; temozolomide; radiation
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Radiotherapy; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ascorbate, radiation, temozolomide (Experimental): Concomitant therapy:
  Radiation therapy, oral temozolomide, and pharmacological ascorbate (ascorbic acid) infusions
  Adjuvant therapy:
  Oral temozolomide and pharmacological ascorbate (ascorbic acid) infusions
  Interventions: Drug: Temozolomide; Radiation: radiation therapy; Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Temozolomide — oral temozolomide (75 mg/m2), given 7 days per week, for a maximum of 49 days during radiation therapy.
  Starting 1 month after radiation therapy, additional temozolomide will be given as chemotherapy cycles. Each cycle is 28 days.
  For the first cycle, temozolomide will be administered (150 mg/m2) once per day for 5 days.
  If the subject tolerates the first cycle well, temozolomide will be prescribed at 200 mg/m2 for cycles 2 through 6. Each cycle is 28 days.
  Other Names: Temodar; Temodal
Radiation: radiation therapy — Conformal radiation administered daily, M-F, to a total dose of 61.2 Gray in 34 fractions.
  Other Names: EBRT; XRT; external beam radiation therapy
Drug: Ascorbic Acid — Intravenous infusions of 87.5g of ascorbate administered three times weekly during radiation.
  After radiation, ascorbate is administered twice weekly through the end of cycle 6 of temozolomide.
  Other Names: Vitamin C; Ascorbate; Pharmacological Ascorbate; 67457-118-50

SUMMARY:
This clinical trial evaluates adding high-dose ascorbate (vitamin C) to standard of care treatment of glioblastoma multiforme (a type of brain tumor) in adults. All subjects will receive high-dose ascorbate in addition to the standard treatment.

DETAILED DESCRIPTION:
Standard treatment for glioblastoma multiforme (GBM) involves maximum safe surgical resection followed by radiation combined with temozolomide (a chemotherapy pill you take by mouth). After radiation, patients receive additional cycles of temozolomide (adjuvant chemotherapy).

Participants will:

* receive high doses of intravenous (IV) ascorbate three times a week during the combined radiation and chemotherapy phase
* receive high doses of intravenous (IV) ascorbate twice a week during adjuvant chemotherapy (after radiation)
* complete health-related quality of life questionnaires pre-radiation, 4 weeks into radiation, 4 weeks after radiation, and then every 3 months. In addition, patients will complete neurocognitive testing pre-radiation, 4 weeks into radiation, 4 weeks after radiation, and approximately 9 months after initiating radiation therapy.

The adjuvant chemotherapy portion of this study lasts for 6 months. After that is completed, participants will go back to standard therapy for their cancer. Participants will continue to have life-long follow-up for this study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign informed consent (power of attorney and/or legally authorized representatives cannot sign on behalf of the patient)
* Patients must have newly diagnosed (i.e., within 5 weeks), histologically or cytologically confirmed glioblastoma multiforme.
* Diagnosis must be made by surgical biopsy or excision.
* Therapy must begin ≤ 5 weeks after surgery or biopsy
* Age ≥ 18 years
* ECOG performance status 0-2. (KPS > 50)
* Absolute neutrophil count (ANC) ≥ 1500 cells per mm3
* Platelets ≥ 100,000 per mm3
* Hemoglobin ≥ 8 g/dL
* Creatinine ≤ 2.0 mg
* Total bilirubin ≤ 1.5 mg/dL
* ALT ≤ 3 times the institutional upper limit of normal
* AST ≤ 3 times the institutional upper limit of normal
* Tolerate one test dose (15g) of ascorbate.
* Not pregnant.

Exclusion Criteria:

* Recurrent high grade glioma
* G6PD (glucose-6-phosphate dehydrogenase) deficiency.
* Patients actively receiving insulin or using a finger-stick glucometer daily for blood glucose measurements
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide.
* Significant co-morbid central nervous system disease, including but not limited to, multiple sclerosis.
* Patients who are on the following drugs and cannot have a drug substitution: warfarin, flecainide, methadone, amphetamines, quinidine, and chlorpropamide.
* Known active concurrent malignancy, as determined by treating physicians.
* Patients who have received prior chemotherapy (including Gliadel wafers) for the current glioma.
* Prior radiation therapy to the head or neck resulting in overlap of RT fields.
* Patients receiving any other investigational agents (imaging agents are acceptable)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection that would result in a hospital stay or delay of treatment, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or impact patient safety.
* Pregnant women.
* Breastfeeding women.
* Known HIV-positive individuals. High-dose ascorbate acid is a known CYP450 3A4 inducer, which results in lower serum levels of antiretroviral drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-03-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | monthly up to 5 years post treatment
  From radiation day 1 until date of death from any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | monthly up to 5 years post treatment
  From radiation day 1 to documented disease progression in MRI imaging as described by the RANO criteria
Adverse Event Frequency | monthly through 7 months post-radiation
  Categorize and quantify using the Common Terminology Criteria for Adverse Events (CTCAE) v. 4 from radiation day 1 through 7 months post-radiation.

OTHER OUTCOMES:
Health-related Quality of Life (HRQOL) | monthly for 3 months, then every 3 months up to 5 years post treatment
  Measure health-related outcomes using the validated EORTC (European Organization for Research and Treatment of Cancer) questionnaires QLQ-C30 and BN-20.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan G. Allen, MD, PhD, Principal Investigator — Assistant Professor, Department of Radiation Oncology, The University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be released publicly as per participant consent and IRB approval. Individual researchers should contact the research team for data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol and informed consent will be shared after primary completion. Statistical analysis plan will be shared with results reporting.
Access Criteria: An IRB-stamped signed usage agreement will be required in addition to a data sharing agreement between the academic centers.

REFERENCES:
- [Background] Schoenfeld JD, Sibenaller ZA, Mapuskar KA, Wagner BA, Cramer-Morales KL, Furqan M, Sandhu S, Carlisle TL, Smith MC, Abu Hejleh T, Berg DJ, Zhang J, Keech J, Parekh KR, Bhatia S, Monga V, Bodeker KL, Ahmann L, Vollstedt S, Brown H, Shanahan Kauffman EP, Schall ME, Hohl RJ, Clamon GH, Greenlee JD, Howard MA, Schultz MK, Smith BJ, Riley DP, Domann FE, Cullen JJ, Buettner GR, Buatti JM, Spitz DR, Allen BG. O2⋅- and H2O2-Mediated Disruption of Fe Metabolism Causes the Differential Susceptibility of NSCLC and GBM Cancer Cells to Pharmacological Ascorbate. Cancer Cell. 2017 Apr 10;31(4):487-500.e8. doi: 10.1016/j.ccell.2017.02.018. Epub 2017 Mar 30. PMID 28366679
- [Derived] Petronek MS, Monga V, Bodeker KL, Kwofie M, Lee CY, Mapuskar KA, Stolwijk JM, Zaher A, Wagner BA, Smith MC, Vollstedt S, Brown H, Chandler ML, Lorack AC, Wulfekuhle JS, Sarkaria JN, Flynn RT, Greenlee JDW, Howard MA, Smith BJ, Jones KA, Buettner GR, Cullen JJ, St-Aubin J, Buatti JM, Magnotta VA, Spitz DR, Allen BG. Magnetic Resonance Imaging of Iron Metabolism with T2* Mapping Predicts an Enhanced Clinical Response to Pharmacologic Ascorbate in Patients with GBM. Clin Cancer Res. 2024 Jan 17;30(2):283-293. doi: 10.1158/1078-0432.CCR-22-3952. PMID 37773633

DOCUMENTS (1):
  • Informed Consent Form (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT02344355/ICF_000.pdf